CLINICAL TRIAL: NCT05893433
Title: Effect of Early Bedside Cycling Exercises on Selected Physical and Psychological Outcomes in Patients After Heart Valve Surgery
Brief Title: Bedside Cycling Exercises Post Heart Valve Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salwa Asem Abusarea Milegy, Teaching assistant in faculty of physical therapy Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cycling valve surgery
Record Dates: First submitted 2023-04-21; First posted 2023-06-07 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient are masked through out the study and health care providers who provide routine care of the patient whether are nurses, physicians or existed physiotherapist are also masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside cycling Group (Experimental): Participants (25 patients) that will receive bedside cycling:
  * Intensity:
    1. RPE from 11 to 13 (scale 6-20)
    2. Resting HR + 20-30 bpm (up to tolerance if non-symptomatic), from low intensity and progressed to medium intensity.
  * Duration: Session duration: Total duration of 20 min, early morning.
  * Frequency: once daily from medically stable until discharge. in addition the medical treatment and routinely physiotherapy protocol.
  Interventions: Device: Bedside cycling
- Routine physical therapy Group (Placebo Comparator): participant that will receive only routine physiotherapy treatment protocol and the medical treatment.
  Interventions: Other: control

INTERVENTIONS:
Device: Bedside cycling — participants receive daily cycling once the patient is relatively stable by weaning off the ventilator and off the require inotropic support and continued to the discharge from the hospital.
  Duration progression if the following conditions are reached:
  1. Initially increase the duration by up to15 min of low exercise time and then increase the intensity after the patient can complete 15- 20 min.
  2. Complete 15min with a medially stable condition gradually until reaching 20 minutes besides the routine physical therapy protocol of breathing exercises, coughing techniques, chest wall vibrations, and mobilization is common during the first postoperative days, The two most frequently used breathing techniques were deep breathing exercises and incentive spirometry and the medical treatment.
  Arms: Bedside cycling Group
Other: control — the routine physical therapy protocol of breathing exercises, coughing techniques, chest wall vibrations, and mobilization is common during the first postoperative days, The two most frequently used breathing techniques were deep breathing exercises and incentive spirometry and the medical treatment.
  Arms: Routine physical therapy Group

SUMMARY:
The aim of this clinical trial is to assess the effect of early bedside cycling exercises post heart valve surgeries. the main question aims to answer: whether adding an early bedside cycling exercise will have an effect on patient's functional capacity, other physical outcomes and have an effect on patient's psychological state?

The participant will be assessed blindly the physical and psychological outcomes before getting randomly allocated in groups. the bedside cycling will be introduced and conducted in the intervention group in addition to the conventional physical therapy cardiac rehabilitation routine through preexisted physical therapy staff who present the hospital:

The routine use of breathing exercises, coughing techniques, chest wall vibrations, and mobilization is common during the first postoperative days.

On the other hand, the control group will only receive the conventional rehabilitation, subsequently, both groups will be assessed and compared by addressing the difference of the outcomes before discharging from the hospital.

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of early bedside cycling exercises on selected physical and psychological outcomes in patients after heart valve surgery.

This study will be carried out on fifty patients diagnosed with valve heart disease and undergoing valve replacement or intervention. They will be recruited from National Heart Institute-Cairo, Egypt.

The purpose, nature and the risk of the study will be explained to the patients and each patient will be consented prior to participation in the study.

The patients in this study will randomly be assigned and randomly allocated into two equal groups (n=25), the intervention group will be treated daily from being extubated and being relatively stable until discharge from the hospital:

* Study group (25 patients): will receive bedside cycling in addition to the medical treatment and physiotherapy protocol.
* Control group (25 patients): will receive only routine physiotherapy treatment protocol and the medical treatment.

The bedside cycling will be introduced and conducted in the intervention group in addition to the conventional phase one of cardiac rehabilitation program through preexisted physical therapy staff who present the hospital.

Bedside cycling: once the patient is relatively stable by weaning off the ventilator and off the require inotropic support and continued until the discharge from the hospital.

* Intensity:

  1. Rating of Perceived exertion scale (RPE) from 11 to 13 (scale 6-20)
  2. post-surgery: resting HR + 20-30 bpm (up to tolerance if non-symptomatic), from low intensity and progressed to medium intensity (According to The American College of Sports Medicine (ASCM) recommendations for prescription of the exercises in phase one of cardiac rehabilitation).
* Duration:

  1. Session duration: Total duration of 20 min, early morning.
  2. Intervention duration: 5-15
  3. Resting as the patient wishes and in case signs of exertion.
  4. Warming up for 5min: low impact, dynamic movement of large group of muscles through available Active Range of Motion (ROM) or introduce to cycling, HR after warming up 10-11 RPE
  5. Cooling down for 5 min or longer: patient observed 30 min after exercise to get to Resting Heart Rate (RHR)
  6. Guided by 11-13 RPE, talk test, 20-30 bpm above RHR (Target HR) and sign and symptoms for stopping exercise. According ASCM recommendations for prescription of the exercises in phase one of cardiac rehabilitation.
* Frequency: once daily from medically stable until discharge.
* Progression if the following conditions are reached:

  1. Initially increase the duration by up to15 min of low exercise time and then increase the intensity after the patient can complete 15- 20 min.
  2. Complete 15min with a medially stable condition
* Precaution:

  1. Vital signs before after and within range
  2. Avoid Valsalva maneuver.

     On the other hand, the control group will only receive the conventional rehabilitation routine:
* The routine use of breathing exercises, coughing techniques, chest wall vibrations, and mobilization is common during the first postoperative days.

Subsequently, both groups will be assessed and compared by addressing the difference of the outcomes before discharging from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty patients with valvular heart disease (VHD)who have undergone valve surgical intervention
2. Their age between 20-40 years old.
3. Both genders

Exclusion Criteria:

1. Cognitive impairment.
2. Neurological disorders.
3. Sever Musculoskeletal disorders (MSD) e.g. (late stages of osteoarthritis).
4. Underlying pulmonary diseases (aspiration pneumonia, chronic obstructive pulmonary disease, pneumothorax, etc).
5. Presence of comorbidities like:

   1. Liver disease e.g. Active cirrhosis or history of previous liver transplant.
   2. Renal disease e.g. Chronic renal disease, Renal failure.
   3. Complicated operative course: post-operative complication:

a) Presence of preoperative cofounder complication: pulmonary hypertension (Pulmonary artery pressure) = which estimated by right ventricular systolic pressure (RVSP) is greater than 50 mmHg, left ventricular dysfunction which estimated left ventricular ejection fraction equals 40 % or less.

b) Patients with Coronary artery bypass surgery, active infective endocarditis, acute valve dysfunction and other acute urgent conditions.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Functional capacity | from the date of patient admission to the hospital until date of the surgical operation, an average of 2 weeks.
  measured by Six Minutes Walk Test, it will be performed on a flat surface, with a predetermined distance 30 meters measured and marked off. Patients will be asked to walk self-paced back and forth between the 2 marked points for 6 minutes. Rests are allowed, and administrators are able to provide standardized feedback during and at the end of the test, The laps are counted, and a distance walked in 6 minutes is determined.
Functional capacity | through study completion, an average of 2 weeks.
  measured by Six Minutes Walk Test, it will be performed on a flat surface, with a predetermined distance 30 meters measured and marked off. Patients will be asked to walk self-paced back and forth between the 2 marked points for 6 minutes. Rests are allowed, and administrators are able to provide standardized feedback during and at the end of the test, The laps are counted, and a distance walked in 6 minutes is determined.
Forced Vital Capacity | from the date of patient admission to the hospital until date of the surgical operation, an average of 2 weeks.
  measured by Spirometry Pulmonary function test, (THOR laboratory Spiro Tube PC Spirometer) will assess Forced Vital Capacity (FCV) in liters.
Forced Vital Capacity | through study completion, an average of 2 weeks.
  measured by Spirometry Pulmonary function test, (THOR laboratory Spiro Tube PC Spirometer) will assess Forced Vital Capacity (FCV) in liters.
Psychological status | from the date of patient admission to the hospital until date of the surgical operation, an average of 2 weeks.
  The Depression Anxiety Stress Scales 42 were used to measure three negative emotional states (depression, anxiety, and stress) experienced by the patients in the previous week. A higher score on the scale indicates a more severe condition, with the highest possible score being 126 and the lowest score being 0.
Psychological status | through study completion, an average of 2 weeks.
  The Depression Anxiety Stress Scales 42 were used to measure three negative emotional states (depression, anxiety, and stress) experienced by the patients in the previous week. A higher score on the scale indicates a more severe condition, with the highest possible score being 126 and the lowest score being 0.
Activities of Daily Living and Functional level | within the first 24-hour post-surgery
  measuring Activities of Daily Living and Function level by using Barthel Index, the current level of 10 items the maximum score is 100, the lower scores ranging from 0- 20 indicating increased disability.
Activities of Daily Living and Functional level | through study completion, an average 7 days
  measuring Activities of Daily Living and Function level by using Barthel Index, the current level of 10 items the maximum score is 100, the lower scores ranging from 0- 20 indicating increased disability.
the Quality of Life | from the date of patient admission to the hospital until date of the surgical operation, an average of 2 weeks.
  The Short Form-12 Health Questionnaire was used to measure the Quality of Life over the past 4 weeks, consisting of two components: physical and mental. The highest possible score for the mental component was 60.75781, indicating a better mental condition. Similarly, the highest possible score for the physical component was 56.577706, indicating a better physical condition.
Length of hospital stay | through study completion, an average of 2 weeks.
  compare the intervention group to control group length of hospital stay.

SECONDARY OUTCOMES:
Functional Capacity | 1 month follow-up.
  measured by Six Minutes Walk Test (6MWT), it will be performed on a flat surface, with a predetermined distance 30 meters measured and marked off. Patients will be asked to walk self-paced back and forth between the 2 marked points for 6 minutes. Rests are allowed, and administrators are able to provide standardized feedback during and at the end of the test, The laps are counted, and a distance walked in 6 minutes is determined.
Psychological status | 1 month follow-up.
  The Depression Anxiety Stress Scales 42 were used to measure three negative emotional states (depression, anxiety, and stress) experienced by the patients in the previous week. A higher score on the scale indicates a more severe condition, with the highest possible score being 126 and the lowest score being 0.
the Quality of Life | 1 month follow-up.
  The Short Form-12 Health Questionnaire was used to measure the Quality of Life over the past 4 weeks, consisting of two components: physical and mental. The highest possible score for the mental component was 60.75781, indicating a better mental condition. Similarly, the highest possible score for the physical component was 56.577706, indicating a better physical condition.
Incidence of adverse event | from the date of beginning cycling intervention or routinely physiotherapy until the date of discharge and will be assessed up to one month.
  the potential incidence of adverse events in both groups will be reported during the study.
Prothrombin International Normalized Ratio (INR) | 1 month follow-up.
  Prothrombin International Normalized Ratio (INR) in the Coagulation profile in both groups will be assessed and provided at one-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Institute (NHI), Giza, Egypt

REFERENCES:
- [Derived] Ahmad AM, Abusarea SA, Fouad BZ, Guirguis SA, Shafie WA. Effect of Adding Early Bedside Cycling to Inpatient Cardiac Rehabilitation on Physical Function and Length of Stay After Heart Valve Surgery: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Jun;105(6):1050-1057. doi: 10.1016/j.apmr.2024.02.711. Epub 2024 Feb 16. PMID 38367831